CLINICAL TRIAL: NCT07024524
Title: Development and Application of A Multimodal Perceptual Evaluation and Precision Rehabilitation System in Congenital Deafness
Brief Title: Perceptual Evaluation and Rehabilitation System Development for Congenital Hearing Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Collaborators: Shanghai Rehabilitation Institute for the Exceptional Children (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2025084-1
Record Dates: First submitted 2025-05-20; First posted 2025-06-17 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Congenital Hearing Loss; Gene Therapy; Speech Perception; Rehabilitation; Reliability and Validity
Keywords: Congenital hearing loss; Gene therapy; Multimodal assessment; Auditory speech perception; Music perception; Spatial hearing; Rehabilitation

STUDY DESIGN:
Intervention Model Description: Stage 1 involved an observational study for reliability and validity assessment, enrolling both healthy subjects and congenital deafness patients . Stage 2 involved an interventional study for rehabilitation training, which included congenital deafness patients .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Congenital Hearing Loss Group (Experimental): The study will recruit patients with congenital hearing loss with hearing thresholds ≥65 dB who have received hearing aids, cochlear implantation, or gene therapy.
  Interventions: Other: Rehabilitation training
- Healthy Controls Group (No Intervention): The study will recruit participants with normal hearing thresholds (≤20 dB) whose age and gender were matched to the patient group.Stage 1 involved an observational study for reliability and validity assessment, enrolling both healthy subjects and congenital deafness patients . Stage 2 involved an interventional study for rehabilitation training, which included congenital deafness patients .Healthy Controls Group were only enrolled in the Stage 1 for reliability and validity assessment, but not the Stage 2 for rehabilitation training.

INTERVENTIONS:
Other: Rehabilitation training — This study constructed a novel multimodal assessment system to evaluate speech perception, music perception, and spatial hearing in congenital deafness patients , and subsequently generated targeted rehabilitation training plan based on the assessment data.
  Arms: Congenital Hearing Loss Group

SUMMARY:
This study aims to establish a novel multimodal evaluation and precision rehabilitation system for patients with congenital hearing loss who have received hearing aids, cochlear implantation, or emerging gene therapy. The proposed system will integrate age-stratified difficulty levels, combined with a gamified interaction platform or software designed to assess and train three core perceptual domains: auditory speech perception, music perception, and spatial hearing capabilities.

DETAILED DESCRIPTION:
For congenital sensorineural hearing loss, the traditional treatment methods are hearing aids and cochlear implantation. In recent years, groundbreaking progress has been made in the field of gene therapy for deafness. However, existing assessment materials and tools are not fully applicable to gene therapy patients. In addition, most assessment materials also show other limitations, including a relatively single assessment dimension with minimal gamified interaction and a lack of age-stratified difficulty levels, etc., which pose challenges in objective and comprehensive evaluation, especially for younger children. There is an urgent need to redesign, optimize, and supplement current assessment tools to more accurately reflect post-treatment multidimensional perceptual function, establish a comprehensive evaluation system, and provide targeted rehabilitation guidance.

Therefore, this study aims to upgrade and develop a novel multimodal evaluation and precision rehabilitation system for patients with congenital hearing loss across different ages and various treatment types. Based on the existing assessment materials and software, the proposed system will combine the gamified method and interactive, friendly interface to construct a set of interesting and interactive measurements, integrating auditory speech, music perception, spatial hearing assessment and rehabilitation training. Patients with congenital hearing loss and healthy controls will be recruited to validate the reliability and validity of the evaluation system and the effectiveness of the rehabilitation training, providing reference for clinical application.

ELIGIBILITY:
Inclusion Criteria:

For Congenital Deafness Group: Patients with congenital hearing loss with hearing thresholds ≥65 dB who have received hearing aids, cochlear implantation, or gene therapy; Age between 1 and 35 years old, regardless of gender.

For Healthy Controls Group: Participants with normal hearing thresholds (≤20 dB) whose age and gender matched to the patient group.

Mandarin Chinese as the native language. Participants and/or their guardians must provide informed consent before the trial, voluntarily sign a written consent form, and commit to receive evaluation at specified time points.

Capable of effective communication with researchers under the guardian's assistance and willing to cooperate and comply with the researchers' requirements.

Participants and/or their guardians should have a correct understanding of the trial and appropriate expectations regarding potential benefits.

Exclusion Criteria:

Presence of other otological disorders that may interfere with the surgical outcome or interpretation of study endpoints, such as otitis media, Meniere's disease, etc.

Presence of other severe congenital diseases, such as congenital heart disease. Presence of severe systemic diseases or in the acute onset of diseases, such as pulmonary tuberculosis, active hepatitis B or C infection, active herpes zoster infection, pancreatitis, renal insufficiency, etc.

Individuals with low immunity, a history of immune deficiency or organ transplantation.

Individuals with a history of neurological, mental disorders, or moderate-to-severe cognitive dysfunction, such as epilepsy, dementia, autism spectrum disorders, etc.

Any other conditions for which the investigators consider the subject unsuitable for participation in this clinical study.

Ages: 1 Year to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-07-04 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-05-05 (Estimated)

PRIMARY OUTCOMES:
Reliability | Baseline
  The reliability of the evaluation system were assessed using Cronbach's α coefficient .
Reliability | Baseline and 1-4 weeks later.
  The test-retest reliability of the evaluation system were assessed using Pearson correlation coefficient.
Validity | Baseline
  The validity of the evaluation system were assessed using Exploratory Factor Analysis, EFA and/or Confirmatory Factor Analysis, CFA.

SECONDARY OUTCOMES:
Effectiveness of the Rehabilitation System | Baseline and 1-3 months after rehabilitation training.
  Changes in the test scores for speech perception from baseline.
Effectiveness of the Rehabilitation System | Baseline and 1-3 months after rehabilitation training.
  Changes in the test scores for music perception from baseline.
Effectiveness of the Rehabilitation System | Baseline and 1-3 months after rehabilitation training.
  Changes in the test scores for spatial hearing perception from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, China